CLINICAL TRIAL: NCT07270822
Title: Implementation of a Systematic Screening for MASLD-related Advanced fibrosiS for Patients With Type 2 Diabetes folLoweD by DIABetologists
Brief Title: Screening for MASLD-related Advanced Fibrosis in Type 2 Diabetes
Acronym: MASLD-DIAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL24_0848
Record Dates: First submitted 2025-09-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Steatotic Liver Disease; Fibrosis of Liver
Keywords: Metabolic dysfunction-associated steatotic liver disease; hepatic transient elastography; hepatic fibrosis; type 2 diabetes mellitus; screening; non-invasive tests
MeSH Terms: conditions — Liver Cirrhosis; Diabetes Mellitus, Type 2 | interventions — Control Groups; Methods

STUDY DESIGN:
Intervention Model Description: Randomized cluster study with two parallel arms:
  * Experimental group: Clusters or private diabetes clinics (five centers) in which a systematic and standardized screening pathway for hepatic AF in patients with T2D has been implemented: calculation of the FIB-4 score and transient elastography measurement performed in diabetes care if FIB-4≥1.30, in accordance with the recommendations of the French Association for the Study of the Liver (AFEF) and the European Association for the Study of the Liver (EASL) .
  * Control group: Clusters or private diabetes practices in which no specific intervention will be deployed (5 centers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative care pathways group (Experimental): Collaborative development of a care pathway for the implementation of a systematic and standardized screening for hepatic AF in patients with T2D in private diabetes clinics.
  The care pathway will include calculation of the FIB-4 score and transient elastography measurement performed in diabetes clinics if FIB-4≥1.30, in accordance with the recommendations of the French Association for the Study of the Liver (AFEF) and the European Association for the Study of the Liver (EASL).
  Interventions: Procedure: Collaborative care pathways group
- Control group without intervention (Other): Current clinical routine practice with no specific intervention
  Interventions: Procedure: Control group without intervention

INTERVENTIONS:
Procedure: Collaborative care pathways group — CO-CONSTRUCTION OF THE CARE PATHWAY:
  Participatory approach according to scientific literature, professional practices, and experience of both healthcare providers and patients.
  Establishment of a working group (hospital endocrinologists, hepatologists, private practice diabetologists, representatives of patients with diabetes followed in the participating centers) to define implementation modalities, professional training, communication and information transfer between professionals, and to ensure a smooth care pathway without overloading the health system .
  IMPLEMENTATION:
  Definition of patient care pathway Training of private diabetologists to integrate FIB-4 and TE measurement into their practices Provision of the FibroScan® Monitoring of patients included in the screening program and of the number of TE measurements performed Validation of TE measurements ≥ 8 kPa in a specialized center Definition of referral procedures for patients towards the specialized center
  Arms: Collaborative care pathways group
Procedure: Control group without intervention — Hepatic AF screening in patients with T2D in private diabetes clinics according to routine care
  Arms: Control group without intervention

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) affects approximately 25% of the global adult population, 25-30% of whom suffer from metabolic dysfunction-associated steatohepatitis (MASH), increasing the risk of progression to advanced fibrosis (AF) (fibrosis stage F3 or cirrhosis F4). Screening for AF is justified because it is associated with an increased risk of overall, hepatic, and cardiovascular mortality and therefore constitutes a public health issue.

Patients with type 2 diabetes (T2D) are identified as a priority target for screening because they are at high risk of AF related to MASLD. The recommendations of the French Association for the Study of the Liver 2020 (afef.asso.fr), the European Association for the Study of the Liver (2024), the American Association of Clinical Endocrinology (2022), and the American Association of Diabetes (2025) all recommend a two-step screening process involving the FIB-4 biological score, followed by transient elastography (TE) if the FIB-4 score is > or = 1.30. Finally, if the TE is ≥8 kPa, the patient is considered to be at intermediate/high risk of AF requiring specialized care to confirm the diagnosis and implement appropriate management, including semi-annual screening for hepatocellular carcinoma in cases of cirrhosis Despite these recommendations, their application in clinical practice remains difficult and requires multidisciplinary collaboration between diabetologists and hepatologists, and between community and hospital sectors, particularly to access TE measures.

Since 2018, the Lyon Sud diabetes department (Hospices Civils de Lyon) has implemented an in-hospital AF screening program using TE for T2D patients. However, this screening by private diabetologists has not yet been implemented, mainly due to the lack of a standardized care pathway and difficulty in accessing TE measurements.

HYPOTHESIS The implementation of systematic and standardized AF screening in private diabetes practices, in two stages and using ET in diabetes care in accordance with recommendations, would significantly increase the identification of patients with AF and thus improve their access to specialized services and appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female
* Type 2 diabetic patient, followed by a diabetologist in private practice participating in the study
* Patient affiliated to a French or European healthcare insurance
* Patient who agrees to be included in the study and who signs the informed consent form

Exclusion Criteria:

* Evidence of advanced fibrosis (F3 or F4 fibrosis based on the results from previous liver biopsy F3 ou F4 or evidence of cirrhosis).
* Evidence of other causes of chronic liver disease
* Patient who does not understand French/ is unable to give consent,
* Patient already included in a trial who may interfere with the study
* The subject is a pregnant or nursing female
* Minor patient
* Patient deprived of liberty,
* Patient admitted to a health or social establishment for purposes other than research
* Mentally unbalanced patients, under supervision or guardianship,
* Patient undergoing psychiatric care
* Patient not affiliated to a healthcare insurance plan
* Patient already included in this screening program in the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1714 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of T2D patients eligible for screening and having undergone AF screening according to the recommendations including assessment of the FIB-4 score, measurement of TE if indicated, and referral for specialized care if required | Between 6 and 12 months following inclusion
  1. Calculation of the FIB-4 score <1.30 (automatic calculation by the medical analysis laboratory or calculated by the liberal diabetologist).
  2. Calculation of the FIB-4 score ≥ 1.30 (automatic calculation by the medical analysis laboratory or calculated by the liberal diabetologist) and realization of a measurement of hepatic TE with either:
     * TE measurement less than 8 kPa OR
     * Measurement of TE greater than or equal to 8kPa and referral for specialized care to a private hepatologist, a hospital hepatology department or the Institute of Hepatology of Lyon at HCL
  According to the recommendations of the EASL (European Association for the Study of the Liver) and the AFEF (French Association for the Study of the Liver), screening includes both the calculation of the FIB-4 score, a transient (TE) measurement, and referral, if indicated, for specialized care.
  ET and FIB-4 measurements cannot be separated

SECONDARY OUTCOMES:
Proportion of patients undergoing transient elastography (TE) measurement | Between 6 and 12 months following inclusion
  measurement among patients with a FIB-4 score ≥ 1.3, as documented in medical records
Proportion of patients referred for specialized consultation for the management of MASLD | Between 6 and 12 months following inclusion
  This include referral to a private hepatologist, a hospital-based hepatology department, or the Hepatology University Hospital Institute (IHU) of Lyon at the Hospices Civils de Lyon (HCL), among those identified through screening
Proportion of patients with TE values ≥ 8 kPa among those referred to specialized care. | Between 6 and 12 months following inclusion
Time interval between successive steps of the screening pathway: FIB-4 assessment, TE measurement, and specialized consultation for the management of MASLD. | Between 6 and 12 months following inclusion
Number of diabetologists not initially participating in implementing the screening pathway (FIB-4 ± TE), | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Statement of discontinuation under study.
Number of patients refusing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Follow-up data
Number of patients eligible for the pathway. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Number of patients included in the care pathway.
Barriers and facilitators to the implementation of the pathway at both individual and organizational levels, as reported by community-based practitioners, specialized care providers and patients. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Interviews with patients
Patient perceptions of their participation in the implementation of the new care pathway | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Interviews with patient's perception of risk, uncertainty, anxiety induced by screening).
Fidelity of the implemented pathway to the predefined specifications, and necessary adaptations. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  % of patients with a compliant care pathway
Transferability of the intervention according to ASTAIRE criteria : characteristics of the target population | Through the inclusion period (after implementation of the new care pathway), an average of 7 months.
  ASTAIRE comprises 23 transferability criteria classified in four categories to analyse the comparability of settings and to facilitate transfer including :
  Category 1 = Typology of the included population : collection and assessment of descriptive data on the population during the initial assessment
Unreliable TE measurements | 2 months after inclusion (strategy implementation period)
  Unreliable TE measurements are defined by IQR/Median ratio ≥0,30. Results will be expressed in number of unreliable measurements
Description of the screening pathway (organization, care trajectory, professional training, patient information and education materials) | 10 months
Proportion of screening compliance among patients with type 2 diabetes (T2D) included in the study (Follow-up period for maintaining the care pathway) | Between 6 and 12 months following inclusion
Number of diabetologists discontinuing participation in the pathway (Follow-up period for maintaining the care pathway) | Between 6 and 12 months following inclusion
Incremental cost-effectiveness ratio (ICER) of implementing a new screening pathway for AF on patients with type 2 diabetes followed in private diabetology practices, compared with usual care | Over a 12-month period
  The outcome measure will be the rate of screenings compliant with the recommendations. The ICER will be interpreted as the additional cost generated by the new screening pathway per additional patient screened
Net budget impact | over a 3-year horizon
  Net budget impact will be assessed in euros for the Mandatory Health Insurance (MHI) at 3 years following the deployment of the new screening strategy for AF in patients with type 2 diabetes managed in private diabetology practices
Transferability according to ASTAIRE criteria: nature of the intervention | Through the inclusion period (after implementation of the new care pathway), an average of 7 months.
  ASTAIRE comprises 23 transferability criteria classified in four categories to analyse the comparability of settings and to facilitate transfer including :
  Category 3 =Typology of the intervention in terms of defining objectives and planning to collect and assess descriptive elements of implementation
Transferability according to ASTAIRE criteria: contextual environment | Through the inclusion period (after implementation of the new care pathway), an average of 7 months.
  ASTAIRE comprises 23 transferability criteria classified in four categories to analyse the comparability of settings and to facilitate transfer including :
  Category 2 = Typology of the environment : collection and assessment of descriptive data on the environment during the initial assessment
Transferability according to ASTAIRE criteria: required implementation strategies. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months.
  ASTAIRE comprises 23 transferability criteria classified in four categories to analyse the comparability of settings and to facilitate transfer including :
  Category 4 = Typology of the implementation strategies required . continuously throughout the project cycle, collect information relating to the terms and conditions of support for the transfer
Inter-observer agreement between measurements performed by diabetologists and by an experienced operator in expert center | Throughout the implementation period up to 2 months after inclusion
  Inter-observer agreement between measurements will explore the procedure for implementing TE in private diabetes clinics. Results will be expressed in percentage of concordant measurements
Single standardized description of the intervention | Throughout the implementation period, an average of 12 months
  The Template for Intervention Description and Replication (TIDIER reporting grid, 12 items, BMJ 2014;348:g1687) will be used. This approach ensures comprehensive and reproducible reporting of all components of the intervention.
Number of diabetologists not initially participating in implementing the screening pathway (FIB-4 ± TE). | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Number of inclusions in the post-implementation phase.
Number of diabetologists not initially participating in implementing the screening pathway (FIB-4 ± TE). | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Percentage of screenings compliant with the recommendations.
Number of patients refusing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Non-realisation of prescribed procedures.
Number of patients refusing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Reasons
Number of patients discontinuing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Follow-up data.
Number of patients discontinuing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Non-realisation of prescribed procedures.
Number of patients discontinuing the screening process | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Reasons
Perceived appropriateness according to community-based and hospital-based professionals. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Professionals' perception of the relevance and alignment of the pathway with their needs (interviews).
Barriers and facilitators to the implementation of the pathway at both individual and organizational levels, as reported by community-based practitioners, specialized care providers and patients. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Interviews with private practitioners.
Barriers and facilitators to the implementation of the pathway at both individual and organizational levels, as reported by community-based practitioners, specialized care providers and patients. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Focus group with specialists from the reference center (diabetologists, endocrinologists, hepatologists)
Fidelity of the implemented pathway to the predefined specifications, and necessary adaptations. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Description of non-compliances
Fidelity of the implemented pathway to the predefined specifications, and necessary adaptations. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Modification of the pathway
Underlying reasons for diabetologists discontinuing participation in the pathway (Follow-up period for maintaining the care pathway) | Between 6 and 12 months following inclusion
Number of diabetologists not implementing the screening pathway (FIB-4 ± TE), and underlying reasons. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Statement of discontinuation under study.
Number of diabetologists not implementing the screening pathway (FIB-4 ± TE), and underlying reasons. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Number of inclusions in the post-implementation phase.
Number of diabetologists not initially participating not implementing the screening pathway (FIB-4 ± TE), and underlying reasons. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Percentage of screenings compliant with the recommendations.
Fidelity of the implemented pathway to the predefined specifications, and necessary adaptations. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Reasons for delays between procedures.
Fidelity of the implemented pathway to the predefined specifications, and necessary adaptations. | Through the inclusion period (after implementation of the new care pathway), an average of 7 months
  Patient-professional and interprofessional relationships within the framework of the care pathway (interviews)
Reasons for diabetologists discontinuing participation in the pathway (Follow-up period for maintaining the care pathway) | Between 6 and 12 months following inclusion

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Diabetology private center, Caluire-et-Cuire
  - Diabetology private center, Lyon
  - Diabetology private center, Saint-Maurice-l'Exil
  - Diabetology private center, Sathonay-Camp